CLINICAL TRIAL: NCT03531853
Title: OCT Technology Development to Assess Ocular Integrity and Characterize Ocular Integrity and Intraocular Scatterers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00092968
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Imaging patients (Experimental): Get uveitis patients and ER patients to image their eyes
  Interventions: Device: hand-held swept source optical coherence tomography

INTERVENTIONS:
Device: hand-held swept source optical coherence tomography — images the eye

SUMMARY:
The purpose of this study is to develop and demonstrate new technologies that will enable a non-contact, compact eye imaging system based on OCT to assist an early responder in acute care settings (like an emergency room) to help assess eye trauma and inflammation (swelling inside the eye).

ELIGIBILITY:
Inclusion Criteria:

- Pre-clinical: employees or students (over the age of 18) of the Duke Eye Center or Biomedical Engineering willing to be imaged with OCT system

- Pilot (ER): patients (over the age of 18) presenting emergently to the Duke Emergency room with traumatic eye injuries and/or suspected open globe

- Pilot (Uveitis): patients presenting to the Duke Eye Center with active uveitis and microhyphema or hyphema; patients who have independently consented to undergo vitreous tap or biopsy for their uveitis care at the Duke Eye Center

Exclusion Criteria:

- Pre-clinical: subject cannot be a direct report to any of the PIs or other key personnel of this study

- Pilot (ER): hemodynamically unstable, unable to consent

- Pilot (Uveitis): unable to consent; cornea or lens opacity/scar which would block the imaging modality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Concordance | Up to 18 months
  By the ability to detect cells in the eye compared to clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kuo, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No